CLINICAL TRIAL: NCT06433661
Title: A Single-centre, Open-label, Randomised, Single-dose, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Etavopivat in Healthy Participants
Brief Title: A Research Study of the Effect of Food on Etavopivat in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN7535-7702; U1111-1289-2544 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers Sickle Cell Disease, Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Etavopivat: fed-fasted (Experimental): Participants will receive a single dose of Etavopivat in fed condition in period 1 and a single dose of Etavopivat in fasted condition in period 2.
  Interventions: Drug: Etavopivat
- Sequence 2: Etavopivat: fasted-fed (Experimental): Participants will receive a single dose of Etavopivat in fasted condition in period 1 and a single dose of Etavopivat in fed condition in period 2.
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — Participants will receive single dose of oral Etavopivat in each treatment period.

SUMMARY:
The purpose of this study is to evaluate the effect of food on the amount of etavopivat in the bloodstream of healthy participants. Participants will take a single oral dose of etavopivat following a high-fat meal (i.e. fed) and on an empty stomach (i.e fasted) on two separate occasions.The study will last up to 50 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 18.5 and 39.9 kilogram per meter square (kg/m^2) (both inclusive) at screening.
* Body weight greater than or equal to (≥) 40.0 kilogram (kg) at screening.
* Considered to be generally healthy based on the medical history, physical examination and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods.
* Participation (i.e., signed informed consent) in any other interventional clinical study within 30 days or 5 times the half-life of the previous investigational medicinal product (IMP) (if known), whichever is longer before screening.
* Any disorder, unwillingness or inability, which in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
* Use of tobacco and nicotine products, defined as any of the below:
* Has used any product containing tobacco or nicotine within 90 days prior to screening,
* Unable or unwilling to refrain from the use of any product containing tobacco or nicotine throughout the study,
* Positive nicotine test at screening.
* Participant is unable to refrain from or anticipates the use of any drug known to be a moderate or strong inhibitor or inducer of uridine 5'-diphospho-glucuronosyltransferase (UGT) enzymes, cytochrome P450 (CYP) 3A4, CYP2C9 or permeability glycoprotein (P-gp), including St. John's Wort, for 28 days prior to dosing and throughout the study.
* Participant is unable to refrain from or anticipate the use of any medications or substances prohibited in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
AUC0-inf, etavopivat: Area under the etavopivat plasma concentration-time curve from 0 hours and extrapolated to infinity after a single dose | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as hours nanograms per milliliter (h*ng/mL).
Cmax, etavopivat: Maximum observed etavopivat plasma concentration after a single dose | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as nanograms per milliliter (ng/mL).

SECONDARY OUTCOMES:
AUC0-last, etavopivat: Area under the etavopivat plasma concentration-time curve from 0 hours to the time of last quantifiable concentration | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as hours nanograms per milliliter (h*ng/ml).
tmax, etavopivat: Time to maximum observed etavopivat plasma concentration after a single dose | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as hours.
t1/2, etavopivat: Terminal half-life for etavopivat after a single dose | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as hours.
CL/Fetavopivat: Apparent plasma clearance of etavopivat after a single dose | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as liter per hours (L/h).
Vz/Fetavopivat: Apparent volume of distribution of etavopivat after a single dose based on plasma concentration values | From 0 to 120 hours after IMP administration (V2/V6)
  Measured as liters (L).
Number of adverse events | From IMP administration on day 1 to completion of the end of study visit (V10)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON-Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com